CLINICAL TRIAL: NCT01078324
Title: Ischemic Colitis Is a Common Cause of Severe Hematochezia and Patient Outcomes Are Worse Than With Other Colonic Diagnoses
Brief Title: Study of Ischemic Colitis Compared to Other Diagnoses in Patients With Lower Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 03-11-115-12; K24DK002650 (NIH)
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Colitis, Ischemic
MeSH Terms: conditions — Colitis, Ischemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ischemic colitis: Ischemic colitis, Diverticulosis

SUMMARY:
The purpose of this study is to study the demographic,laboratory,endoscopic, and outcomes of ischemic colitis patient presented with severe lower gastrointestinal bleeding compared to other diagnoses.

DETAILED DESCRIPTION:
Secondary purpose of this study is to assess the risk factors for predicting diverticulosis versus ischemic colitis.

ELIGIBILITY:
Inclusion Criteria:

* bright red blood clots or burgundy colored stool documented by a health care worker
* clinical or laboratory evidence of significant blood loss, manifested by any one of the following: (a) more than three bloody bowel movements in eight hours (b) a decrease of two grams of hemoglobin (Hgb) from baseline, or (c) transfusion of more than three units of red blood cell (URBC).

Exclusion Criteria:

* age less than 18 year
* history of inflammatory bowel disease
* hypotension or shock refractory to resuscitation
* severe coagulopathy refractory to resuscitation (platelet count < 30,000; prothrombin time [PT]- more than 2 times normal; partial thromboplastin time [PTT]- more than 2 times normal)
* acquired immune deficiency syndrome or neutropenia
* the inability to provide informed consent
* documentation of anal disorders as a cause of bleeding such as internal hemorrhoids, anal fissures, polyps or cancer of the anal canal, and fistulae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted into the hospital
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 1997-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The clinical course and outcomes of the ischemic colitis group compared to other colonic diagnoses group | 12 year period

SECONDARY OUTCOMES:
Risk factors and prediction of ischemic colitis versus diverticulosis as the cause of severe hematochezia | 12 year period

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Jensen, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- The Veterans Affairs Greater Los Angeles Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Jensen DM, Machicado GA. Diagnosis and treatment of severe hematochezia. The role of urgent colonoscopy after purge. Gastroenterology. 1988 Dec;95(6):1569-74. doi: 10.1016/s0016-5085(88)80079-9. PMID 3263294
- [Background] Jensen DM, Machicado GA. Colonoscopy for diagnosis and treatment of severe lower gastrointestinal bleeding. Routine outcomes and cost analysis. Gastrointest Endosc Clin N Am. 1997 Jul;7(3):477-98. PMID 9177148
- [Background] Jensen DM, Machicado GA, Jutabha R, Kovacs TO. Urgent colonoscopy for the diagnosis and treatment of severe diverticular hemorrhage. N Engl J Med. 2000 Jan 13;342(2):78-82. doi: 10.1056/NEJM200001133420202. PMID 10631275